CLINICAL TRIAL: NCT01786499
Title: The Effect of Relaxation Response on Provider Burnout
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 3888-2
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Burnout; Resilience; Perceived Stress
Keywords: Burnout; Stress; Provider; Relaxation Response
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Relaxation Response Training (Other)
  Interventions: Behavioral: Relaxation Response Training

INTERVENTIONS:
Behavioral: Relaxation Response Training

SUMMARY:
Hypothesis: Relaxation Response training is an effective intervention in reducing the prevalence and severity of burnout and its components from baseline levels among physicians receiving the training intervention. The intervention is hypothesized to moderate the relationship between Areas of Worklife (AWS) and burnout by improving physician's ability to cope with the demands of their workplace. This increased coping ability is hypothesized to reduce burnout.

Physician practices are as unique as the individual practitioners and the environment in which they practice. Traditional instruction of relaxation or self-care techniques has required participants to travel to locations remote from the workplace. The time commitment required for this behavior is additive to the time required to learn the intervention and of itself may induce extra stress increasing the potential for burnout. This study proposes that bringing the intervention to the workplace will increase provider willingness to participate and diminish the stress introduced by deployment of the intervention. Since inpatient and outpatient medicine have different practice characteristics and demands on the time of the practitioners, this study will need to develop and test the logistics necessary to bring the training to the different physician populations.

ELIGIBILITY:
Inclusion Criteria:

* Providers at designated clinic and hospital

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in burnout expression in study population | Three months
  Measurement strategy: data collection at Baseline (prior to beginning of the Relaxation Response training), 3 months, 6 months, 12 months, 18 months, and 24 months after implementation.
  Measurement instruments: survey that measures prevalence and severity of burnout (Maslach Burnout Inventory, MBI), the proximate drivers of burnout (Areas of Worklife Survey), an assessment of the perceived stress experienced by the practitioners (Perceived Stress Scale), and a measure of the personal resilience (Conor-Davidson Resilience Scale). Standard univariate statistics will be used to produce descriptive measures of the sample, Chronbach's alpha to assess internal reliability of survey measures, and confirmatory factor analysis will be employed to determine if the data fits the a priori theoretical model. A combination of the approaches above will help to assess the effectiveness of the Relaxation Response intervention on the prevalence, incidence, and trajectory of provider burnout.

CONTACTS AND LOCATIONS:
Locations (1):
- Allina Health, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Benson H, Greenwood MM, Klemchuk H. The relaxation response: psychophysiologic aspects and clinical applications. Int J Psychiatry Med. 1975;6(1-2):87-98. doi: 10.2190/376W-E4MT-QM6Q-H0UM. PMID 773864
- [Background] Leiter, M. P., & Maslach, C. (2004). Areas of worklife: A structured approach to organizational predictors of job burnout. Research in Occupational Stress and Well being: Emotional and Physiological Processes and Positive Intervention Strategies, 3, 92-134.